CLINICAL TRIAL: NCT04634266
Title: TRICuspid Intervention in Heart Failure Trial (TRICI-HF-DZHK24)
Brief Title: TRICuspid Intervention in Heart Failure Trial
Acronym: TRICI-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LMU Klinikum (Other)
Collaborators: Heart and Diabetes Center North Rhine-Westphalia (Other); University Medical Center Mainz (Other); Heart Center Leipzig - University Hospital (Other); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); University of Leipzig (Other)
Responsible Party: Principal Investigator, Thomas Stocker, MD, LMU Klinikum
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TRICI-HF; TRICI-HF-DZHK24 (Other Grant/Funding Number: Deutsches Zentrum für Herzkreislaufforschung)
Record Dates: First submitted 2020-11-17; First posted 2020-11-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure Attributable to Severe Tricuspid Regurgitation

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, multicenter, randomized, open label trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention (Experimental): Transcatheter tricuspid valve treatment (TTVT) plus optimal medical therapy (OMT)
  Interventions: Device: Transcatheter tricuspid valve treatment (TTVT)
- Control intervention (No Intervention): OMT for severe tricuspid regurgitation in right-sided heart failure

INTERVENTIONS:
Device: Transcatheter tricuspid valve treatment (TTVT) — Percutaneous CE-mark approved techniques for transcatheter tricuspid valve treatment (TTVT): These include (I) transcatheter annuloplasty devices (Tricuspid Cardioband) and (II) transcatheter edge-to-edge repair (TriClip, PASCAL).
  Arms: Experimental intervention

SUMMARY:
Functional tricuspid regurgitation (TR) is a serious and progressive disease. Guidelines recommend surgical valve repair of severe TR in symptomatic patients. Despite its association with excess mortality and morbidity, TR has been relatively neglected and is severely undertreated. In particular this is because isolated tricuspid surgery remains associated with high mortality rates, and thus, patients with severe TR are often deemed inoperable due to severe co-morbidities and frailty. In recent years, percutaneous CE-mark approved techniques for transcatheter tricuspid valve treatment (TTVT) have emerged as alternatives to surgery. These include (I) transcatheter annuloplasty devices (Tricuspid Cardioband) and (II) transcatheter edge-to-edge repair (TriClip, PASCAL). Several non-randomized studies suggested improved functional outcomes after TTVT, however, to data there is no evidence from randomized controlled trials addressing the actual efficacy of TTVT. The TRICuspid Intervention in Heart Failure trial (TRICI-HF trial) will assess the concept that TTVT will translate into a reduced morbidity and mortality. Patients will be randomly assigned in a 2:1 fashion to TTVT plus OMT (Experimental group) or OMT alone (Control group). TRICI-HF is an industry-independent, investigator-initiated strategy study and investigators may choose any suitable CE-marked percutaneous system "on-label" for TTVT.

ELIGIBILITY:
The following inclusion criteria were defined to assure generalizability of the population to be studied:

* Subject is symptomatic due to severe TR despite being on stable OMT for at least 30 days based on judgment of the local heart team. Patients with reduced left ventricular ejection fraction (HFrEF) will likely constitute a minority among eligible patients with isolated severe tricuspid regurgitation (9,13). However, HFrEF patients enrolled into the trial need to be on stable guideline-directed medical therapy for at least 4 weeks..
* Subject is at intermediate or greater estimated risk of mortality with tricuspid valve surgery based on judgment of the local heart team
* New York Heart Association (NYHA) Functional Class II, III or IVa
* Femoral vein access and valve anatomy are determined to be feasible for interventional treatment (including sufficient quality of TTE and TEE imaging)
* Age ≥ 18 years at time of consent
* Subject must provide written informed consent prior to any trial related procedure

The following exclusion criteria were selected to define a representative study cohort:

* Presence of severe aortic, mitral or pulmonary valve disease OR surgical/interventional treatment at the aortic, mitral or pulmonary valves prior 60 days
* Right heart catheterization (mandatory) with systolic pulmonary artery pressure > 70 mmHg or substantial pre-capillary pulmonary hypertension (defined as mean pulmonary artery pressure (mPAP) >30 mmHg plus transpulmonary gradient (TPG) >17 mmHg or pulmonary vascular resistance (PVR) >5 wood units)
* Tricuspid valve stenosis (tricuspid mean gradient > 5 mmHg)
* Pacemaker or ICD leads that would prevent appropriate TTVT
* Prior tricuspid valve procedures or tricuspid valve leaflet anatomy that would interfere with appropriate TTVT (e.g. calcification, Ebstein anomaly, coaptation defect > 8mm for planned leaflet- and annuloplasty-based therapy)
* Chronic renal failure requiring dialysis
* Tricuspid valve anatomy not evaluable by TTE and TEE
* Myocardial infarction or cerebrovascular accident within prior 90 days
* Life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality or heart failure hospitalization | 12 months
  Composite of time to all-cause mortality or heart failure hospitalization - whichever occurs first - at a minimum follow-up of 12 months

SECONDARY OUTCOMES:
All-cause mortality (unadjusted and adjusted for TR severity at baseline) | 12 months
Heart failure hospitalizations (frequency and length; unadjusted and adjusted for TR severity at baseline) | 12 months
Change in Quality of Life as assessed by the MLHFQ from baseline | 12 months
Re-intervention rates for recurrent tricuspid regurgitation | 12 months
Change in NYHA Class from baseline (≥III/IV to ≤I/II) | 12 months
Change in 6 minute walk test distance from baseline | 12 months
Change in echocardiographic parameters (among others: TR grade I-V, RV dimension and function, LV dimension and function, estimation of sPAP) | 12 months
Development of tricuspid stenosis (mean inflow gradient >5mmHg) | 12 months
Change in peripheral edema assessed by the edema scale (grade I-IV) and subject weight (kilograms) from baseline | 12 months
Change of diuretic drugs and heart failure medications from baseline (type and dosage) | 12 months
Change in laboratory markers for cardiac, renal and hepatic function (complete blood count, NT-proBNP, eGFR, serum creatinine, bilirubin, AST, ALT and gGT) | 12 months

OTHER OUTCOMES:
Safety of transcatheter tricuspid valve intervention | 1 month
  Major adverse events that are related to the intervention and are relevant for patients undergoing TTVT: Mortality, life threatening bleeding (defined as BARC bleeding type 3 and 5), major vascular or cardiac structural complications requiring intervention, or mechanical circulatory support.

CONTACTS AND LOCATIONS:
Locations (23):
- Germany (23):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Schüchtermann-Klinik, Bad Rothenfelde
  - Charité Universitätsmedizin Berlin, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Herzzentrum Uniklinik Köln, Cologne
  - St.-Johannes-Hospital Dortmund, Dortmund
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Giessen, Giessen
  - Herzzentrum Göttingen, Göttingen
  - Herzzentrum UKE, Hamburg
  - Katholisches Marienkrankenhaus Hamburg, Hamburg
  - MVZ Prof. Mathey/Schofer, Hamburg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Herzentrum Leipzig, Leipzig
  - Universitätsmedizin Mainz, Mainz
  - LMU Klinikum, München
  - Herzzentrum Siegburg, Siegburg

IPD SHARING:
Plan to Share IPD: Undecided